CLINICAL TRIAL: NCT06155669
Title: The Impact of Virtual Reality -Guided Visual and Auditory Therapy on Symptom Severity and Psychological Well-Being in Tension-Type Headache Patients: A Controlled Study
Brief Title: The Use of Virtual Reality Applications in Tension-Type Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Virtual Reality Tension Type
Record Dates: First submitted 2023-11-26; First posted 2023-12-04 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Headache; Analgesia; Tension-Type Headache
MeSH Terms: conditions — Headache; Agnosia; Tension-Type Headache

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standart Group (No Intervention): Participants will be selected from patients diagnosed with tension-type headache according to the International Classification of Headache Disorders, third edition (ICHD-3) criteria. All selected participants will be administered 25 mg of dexketoprofen.
- Virtual Reality (Experimental): Participants will be selected from patients diagnosed with tension-type headache according to the International Classification of Headache Disorders, third edition (ICHD-3) criteria. Selected participants, in addition to being administered 25 mg of dexketoprofen, will also use virtual reality goggles.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Participants will be selected from patients diagnosed with tension-type headache according to the International Classification of Headache Disorders, third edition (ICHD-3) criteria. Selected participants, in addition to being administered 25 mg of dexketoprofen, will also use virtual reality goggles.
  Arms: Virtual Reality

SUMMARY:
The primary aim of this research is to objectively assess the impact of virtual reality (VR) technology on pain symptoms in tension-type headache patients. This study is designed to understand the potential of VR in the treatment of tension-type headaches, exploring its ability to reduce pain severity and improve patients' quality of life.

DETAILED DESCRIPTION:
Tension-type headache is a prevalent health issue that can cause significant discomfort to patients. The potential use of VR goggles as an effective alternative treatment option in these patients is crucial in clinical applications. The quality of life of tension-type headache patients is often affected. If VR goggle technology can enhance the quality of life for these patients, it would be a significant finding.

Additionally, our research may contribute more data to the scientific literature on the impact of VR goggle technology in headache treatment. This could assist future researchers in designing similar studies and better understanding the results. If VR goggle technology proves effective, it could contribute to diversifying treatment options for tension-type headache patients and improving access to treatment.

The primary objective of the study is to investigate the effect of virtual reality therapy on pain symptoms in tension-type headache patients. If the results are positive, VR technologies may alleviate pain and enhance the quality of life for these patients. It could also help them function better in their daily lives. If relaxation is found to be effective in the VR group, a new treatment option would be introduced for tension-type headache patients. This could contribute to the diversification of treatment options.

The study poses no risk to the patient. The patient will lie on the bed, and the VR goggles will be used accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 65
* Patients meeting the criteria for Tension-Type Headache (TTH) in the third edition of the International Classification of Headache Disorders
* Patients willing to participate in the study
* Patients indicating a VAS score of 50 and above
* Patients without other suspected diagnoses
* Patients with no known history of adverse reactions to the active ingredients of the drugs to be used
* Conscious patients
* Patients who are oriented and cooperative

Exclusion Criteria:

* Patients under the age of 18 and over the age of 65
* Patients who do not consent to participate in the study
* Patients with vital signs outside normal limits
* Patients with a history of adverse reactions to known NSAIDs
* Individuals unable to determine pain intensity on the VAS
* Patients with a VAS score of 50 mm and below
* Pregnant individuals
* Those with advanced systemic diseases
* Patients with malignancies
* Individuals with chronic liver and kidney diseases
* Those using sedative and analgesic neuro-psychiatric drugs
* Individuals with a history of psychological and neurological diseases
* Patients who used analgesics within 8 hours before the examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in Pain Intensity Measured by Visual Analog Skala (VAS) | Baseline (VAS-0) to 30th, 60th, and 120th minutes post-treatment.
  Change in pain intensity was assessed using the Visual Analog Scale (VAS), where participants rated their pain on a scale from 0 mm (no pain) to 100 mm (worst pain ever experienced). The primary outcome was the change in VAS scores from baseline (VAS-0) to subsequent time points (VAS-30, VAS-60, and VAS-120), calculated as ΔVAS and ΔVAS% for each interval.

SECONDARY OUTCOMES:
Mood Improvement Measured by Likert Scale | Baseline to the 120th minute post-treatment.
  Participants' mood was assessed using a 5-point Likert scale, ranging from 1 (Very Poor) to 5 (Very Good). Mood scores were evaluated at baseline (Likert-0) and at the 120th minute (Likert-120), with the difference used to determine changes in mood.
Occurrence of Side Effects | From baseline to the 120th minute post-treatment.
  Side effects, including dizziness, nausea, or other symptoms, were recorded through patient self-reports and observations by research staff at the 30th, 60th, and 120th minutes.

CONTACTS AND LOCATIONS:
Overall Officials: SAFA DÖNMEZ, M.D., Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashina S, Mitsikostas DD, Lee MJ, Yamani N, Wang SJ, Messina R, Ashina H, Buse DC, Pozo-Rosich P, Jensen RH, Diener HC, Lipton RB. Tension-type headache. Nat Rev Dis Primers. 2021 Mar 25;7(1):24. doi: 10.1038/s41572-021-00257-2. PMID 33767185
- [Result] Almedhesh SA, Elgzar WT, Ibrahim HA, Osman HA. The effect of virtual reality on anxiety, stress, and hemodynamic parameters during cesarean section: A randomized controlled clinical trial. Saudi Med J. 2022 Apr;43(4):360-369. doi: 10.15537/smj.2022.43.4.20210921. PMID 35414614
- [Result] Bagher SM, Felemban OM, Alandijani AA, Tashkandi MM, Bhadila GY, Bagher AM. The effect of virtual reality distraction on anxiety level during dental treatment among anxious pediatric patients: a randomized clinical trial. J Clin Pediatr Dent. 2023 Jul;47(4):63-71. doi: 10.22514/jocpd.2023.036. Epub 2023 Jul 3. PMID 37408348
- [Result] Loder E, Rizzoli P. Tension-type headache. BMJ. 2008 Jan 12;336(7635):88-92. doi: 10.1136/bmj.39412.705868.AD. No abstract available. PMID 18187725
- [Result] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Result] Burch R. Migraine and Tension-Type Headache: Diagnosis and Treatment. Med Clin North Am. 2019 Mar;103(2):215-233. doi: 10.1016/j.mcna.2018.10.003. Epub 2018 Dec 3. PMID 30704678
- [Result] Yavuz E, Gulacti U, Lok U, Turgut K. Intravenous metoclopramide versus dexketoprofen trometamol versus metoclopramide+ dexketoprofen trometamol in acute migraine attack in the emergency department: A randomized double-blind controlled trial. Am J Emerg Med. 2020 Nov;38(11):2254-2258. doi: 10.1016/j.ajem.2020.04.038. Epub 2020 Apr 15. PMID 32359776